CLINICAL TRIAL: NCT02741141
Title: A Comparative Study of the Effect of Two Partographs on the Cesarean Section Rate in Women in Spontaneous Labour
Acronym: PARTODYS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the study was stopped due to a change in delivery room practices
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 6225
Record Dates: First submitted 2016-01-12; First posted 2016-04-18 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Dystocia
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Classical partograph (Active Comparator): Labour dystocia is diagnosed when cervical dilation is less than 1 cm per hour or after 3 hours at complete cervical dilation without engagement of the presentation. In this case, active management of labour is started with introduction of oxytocin, artificial rupture of membranes and supportive therapy.
  Interventions: Other: Classical partograph
- New partograph (Experimental): The second strategy is based on the partograph developped by Neal and Lowe. An active management of labour is started when crossing the dystocia line or when there are no cervical modifications after 4 hours beyond 5 cm of cervical dilation. In this case, active management of labour is started with introduction of oxytocin, artificial rupture of membranes and supportive therapy.
  Interventions: Other: New partograph based on the studies of Neal and Lowe

INTERVENTIONS:
Other: New partograph based on the studies of Neal and Lowe — The partograph designed by Neal and Lowe includes an "action line" which if crossed permits an active management of labour.
  Eventually, the only difference between the two arms is the moment when the active management of labour is started.
  The oxytocin is administrated according to the department protocol.
  Arms: New partograph
Other: Classical partograph — Classical partograph used as standard care
  Arms: Classical partograph

SUMMARY:
In the 2010-french perinatal survey, the overall cesarean section (CS) rate during labour was 21 % and 16% to 38% in case of dystocia.

The definition of " dystocia " is traditionally based on the research led by Friedman in the 1950's on a restricted population sample. Several studies over the last years seem to indicate that the different phases of labour are longer than originally described by Friedman.

Our current hypothesis is that the application of a new definition of dystocia would enable a more appropriate management of labour.

DETAILED DESCRIPTION:
The main purpose of this study is to show a significant decrease of the CS rate with the use of the new partograph developed by Neal and Lowe.

Secondary purposes are

* To reduce the use of oxytocin during labour without increasing maternal or neonatal morbidity;
* To decrease immediate per-operative complications and post-operative complications associated with CS

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

* Affiliation to a social security insurance
* Written consent given
* Singleton pregnancy
* Cephalic presentation
* ≥37 gestational weeks
* Spontaneous onset of labour

Exclusion Criteria:

* Previous cesarean section
* Induction of labour
* Intrauterine growth restriction
* In utero fetal death
* Congenital malformation
* Chorioamnionitis
* Placenta praevia
* Need for an emergency delivery (fetal heart rate abnormalities at admission)
* Contra-indication for vaginal delivery
* Patient under temporary guardianship, guardianship or judicial protection
* Patient included in another study which could interfere with the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 633 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Cesarean section rate (all causes) | From admission in the labour ward to the delivery (duration from 0 to 24 hours approximately)

SECONDARY OUTCOMES:
obstetrical measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Total amount of oxytocin used (mUI)
obstetrical measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Rate of uterine hyperstimulation (%)
obstetrical measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Rate of post-partum hemorrhage (%)
obstetrical measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Rate of uterine rupture (%)
obstetrical measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Rate of retained placenta (%)
obstetrical measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Need of an artificial rupture of membranes (Y/N)
obstetrical measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Color of the amniotic fluid
obstetrical measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Duration of the first and second stages of labour
obstetrical measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Rate of vaginal delivery (spontaneous or assisted) (%)
obstetrical measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Rate of cesarean section (according to indication) (%)
Maternal measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Need for an epidural or general anaesthesia
Maternal measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Transfusion rate (%)
Maternal measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Maternal fever during labour (°C)
Maternal measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Rate of thrombo-embolic events (%)
Maternal measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Rate of third- and fourth-degree perineal tears and episiotomy (%)
Maternal measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Rate of surgical site infection, endometritis or septicemia (%)
Neonatal measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Neonatal arterial umbilical cord pH < 7,00 and/or BD > 12 mmol/L
Neonatal measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Apgar score < 7 at 5 minutes
Neonatal measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Transfer to intensive care unit rate
Neonatal measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Neonatal infection rate (%)
Neonatal measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Neonatal convulsion rate (%)
Neonatal measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Rate of neonatal deaths (%)
Neonatal measures associated with possible effects of both strategies on maternal and fetal outcome | From the admission in the labour ward until the dismissal from maternity (2 to 5 days)
  Neonatal encephalopathy rate (or the introduction of therapeutic hypothermia)

CONTACTS AND LOCATIONS:
Overall Officials: Adrien GAUDINEAU, Principal Investigator — Strasbourg's University Hospitals
Locations (1):
- University Strasbourg Hospital, Strasbourg, France